CLINICAL TRIAL: NCT07170696
Title: The Impact of Dialogic Reading-Based Nutrition Education on Preschool Children's Nutrition Knowledge and Dietary Diversity: A Quasi-Experimental Study
Brief Title: Dialogic Reading-Based Nutrition Education on Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Müberra DEMİRBAŞ, Research Assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/6
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Nutrition Knowledge; Dietary Diversity
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dialogic Reading-Based Nutrition Education (Experimental): The intervention group received an eight-week nutrition education program that integrated dialogic reading with real food exposure, sensory play, table-top activities, and parental involvement.
  Interventions: Behavioral: nutrition education
- Control group (No Intervention): No intervention was applied to the control group

INTERVENTIONS:
Behavioral: nutrition education — dialogic reading-based nutrition education
  Arms: Dialogic Reading-Based Nutrition Education

SUMMARY:
This study aims to evaluate the effectiveness of a dialogic reading-based nutrition education program in improving nutrition knowledge and dietary diversity among preschool children.

DETAILED DESCRIPTION:
This study uses a quasi-experimental pre-test-post-test design. A total of 46 children (26 in the intervention group and 20 in the control group) from two preschools in Istanbul are included. The intervention group receives an eight-week nutrition education program that integrates dialogic reading with real food exposure, sensory play, table-top activities, and parental involvement.

Data are collected using the Children Nutrition Knowledge Form, Dietary Diversity Scale, and anthropometric measurements. The study is designed to assess whether a dialogic reading-based and multi-component nutrition education program can enhance preschool children's nutrition knowledge and dietary diversity.

ELIGIBILITY:
Inclusion Criteria:

* Parental consent for participation
* Regular school attendance
* No medical condition requiring a special diet
* No diagnosis of congenital or acquired developmental delay/disability
* No prior participation in a nutrition-focused developmental support program

Exclusion Criteria:

* Special needs
* Missing family form
* Foreign language (not fluent in study language)
* Absenteeism

Ages: 60 Months to 66 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2024-10-09 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
nutrition knowledge | From enrollment to the end of treatment at 8 weeks
  The Child Nutrition Knowledge Form is based on the "Eat Smart with MyPyramid for Kids" educational material developed by the United States Department of Agriculture. The Turkish adaptation of the form was conducted by Başkale in 2010. The form includes images of 30 food items from five food groups and consists of five questions. It is administered face-to-face with preschool children by reading each question aloud and asking the child to indicate the correct answer by pointing to the relevant image. Each correct answer is scored as 1, and incorrect answers are scored as 0. Therefore, the total possible score ranges from 0 to 20. A higher score indicates a higher level of nutrition knowledge .
dietary diversity | From enrollment to the end of treatment at 8 weeks
  The Dietary Diversity Score was calculated based on the Food and Agriculture Organization (FAO) Dietary Diversity Questionnaire . A non-quantitative food frequency questionnaire was used to assess the frequency of consumption of eight food groups (dairy products, fresh meats, eggs, fish and seafood, legumes, nuts and seeds, vegetables, fruits, and cereals). If the consumption frequency of any food in these groups was marked as "Every day," "3-5 times a week," or "1-2 times a week," 1 point was assigned. If it was marked as "Once every 15 days," "Once a month," "Rarely," or "Never," 0 points were assigned.

CONTACTS AND LOCATIONS:
Overall Officials: Asya Evci, Study Chair — Istanbul Medeniyet University
Locations (1):
- Müberra Demirbaş, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz-Onal H, Demirbas M, Edis-Karaman M, Evci-Guney SA. The impact of dialogic reading-based nutrition education on preschool children's nutrition knowledge and dietary diversity: a quasi-experimental study. BMC Public Health. 2025 Dec 2;26(1):83. doi: 10.1186/s12889-025-25792-5. PMID 41331874